CLINICAL TRIAL: NCT04695977
Title: A Randomized, Open-label, Active-control, Phase 2/3 Study of First-line Intratumoral CMP-001 in Combination With Intravenous Nivolumab Compared to Nivolumab Monotherapy in Subjects With Unresectable or Metastatic Melanoma
Brief Title: CMP-001 in Combination With Nivolumab Compared to Nivolumab Monotherapy in Subjects With Advanced Melanoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-011
Record Dates: First submitted 2020-12-10; First posted 2021-01-06 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Advanced Melanoma; Metastatic Melanoma; Unresectable Melanoma
Keywords: vidutolimod
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CMP-001 and Nivolumab (Experimental): All enrolled subjects will receive CMP-001 IT and nivolumab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: CMP-001; Drug: Nivolumab
- Nivolumab Monotherapy (Experimental): All enrolled subjects will receive nivolumab monotherapy IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: CMP-001 — Subjects will receive CMP-001 10 mg IT weekly for 7 doses after which CMP-001 will be administered every 3 weeks (Q3W).
  Other Names: vidutolimod
  Arms: CMP-001 and Nivolumab
Drug: Nivolumab — Nivolumab 360 mg IV is administered Q3W.
  Other Names: OPDIVO

SUMMARY:
CMP-001-011 is a Phase 2/3 study of CMP-001 intratumoral (IT) and nivolumab intravenous (IV) compared to nivolumab monotherapy administered to participants with unresectable or metastatic melanoma.

The study is divided into two phases: Phase 2 and Phase 3.

The primary objective of Phase 2 of the study is to determine confirmed objective response rate (ORR) for treatment with first-line CMP-001 in combination with nivolumab versus nivolumab monotherapy in subjects with unresectable or metastatic melanoma.

The secondary objective of Phase 2 of the study is to evaluate the safety and tolerability of first-line CMP-001 in combination with nivolumab versus nivolumab monotherapy in subjects with unresectable or metastatic melanoma.

The primary objective of Phase 3 of the study is to evaluate progression-free survival (PFS) for subjects receiving first-line CMP-001 in combination with nivolumab versus nivolumab monotherapy for unresectable or metastatic melanoma.

The secondary objectives of Phase 3 are to:

* To evaluate the safety and tolerability of first-line CMP-001 in combination with nivolumab versus nivolumab monotherapy in subjects with unresectable or metastatic melanoma.
* To evaluate the efficacy of first-line CMP-001 in combination with nivolumab versus nivolumab monotherapy in subjects with unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study must meet all of the following inclusion criteria to be eligible:

1. Histologically or cytologically confirmed unresectable Stage III or Stage IV melanoma per AJCC Cancer Staging Manual Eighth Edition.
2. Measurable disease, as defined by RECIST v1.1 and both of the following:

   1. At least 1 accessible lesion amenable to repeated IT injection
   2. One or more measurable lesions at least 1 cm in diameter that are not intended for CMP-001 injection and can be followed as target lesions per RECIST v1.1
3. Able to provide tissue from a core or excisional biopsy (fine needle aspirate is not sufficient). A newly obtained biopsy (within 90 days before the first dose of study treatment) is preferred, but an archival sample is acceptable if no intervening therapy for melanoma/cancer was received. Note: for tissue sampling details, please refer to the Laboratory Manual.
4. Adequate organ function based on most recent laboratory values within 3 weeks before the first dose of study treatment on Week 1 Day 1 (W1D1):

   1. Bone marrow function:

      * neutrophil count ≥1500/mm3
      * platelet count ≥ 100 000/mm3
      * hemoglobin concentration ≥9 g/dL
      * white blood cells ≥2000/mm3
   2. Liver function:

      * total bilirubin ≤1.5 × the upper limit of normal (ULN) with the following exception: subjects with Gilbert Disease total serum bilirubin ≤3 × ULN
      * aspartate aminotransferase and alanine aminotransferase ≤3 ×ULN
   3. Lactate dehydrogenase ≤2 × ULN
   4. Renal function: estimated (Cockcroft-Gault) or measured creatinine clearance ≥30 mL/min
   5. Coagulation

      * International normalized ratio or prothrombin time (PT) ≤ 1.5 × ULN, unless subject is receiving anticoagulant therapy, as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
      * Activated partial thromboplastin time or PTT ≤1.5 × ULN, unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
5. Eastern Cooperative Oncology Group Performance Status of 0 to 1 at Screening.
6. Age ≥18 years at time of consent.
7. Capable of understanding and complying with protocol requirements.
8. Women of childbearing potential must have negative serum pregnancy test prior to dosing at W1D1 and be willing to use an adequate method of contraception from the time of consent until at least 150 days after the last dose of study treatment.
9. Male subjects must be surgically sterile or must agree to use adequate method of contraception from the time of consent until at least 210 days after the last dose of study treatment.
10. Able and willing to provide written informed consent and to follow study instructions.

Subjects unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

Subjects presenting with any of the following will not qualify for entry into the study:

1. Uveal, acral, or mucosal melanoma.
2. Received prior systemic treatment for melanoma in the unresectable or metastatic setting. Prior adjuvant therapy is acceptable if the treatment course (of approximately 1 year duration) was completed and there was no recurrence within 6 months of the last dose of adjuvant treatment.
3. Received prior therapy with CMP-001.
4. Requires systemic pharmacologic doses of corticosteroids greater than the equivalent of 10 mg/day prednisone within 30 days before the first dose of study treatment on W1D1.

   1. Subjects who are currently receiving steroids at a prednisone-equivalent dose of ≤10 mg/day do not need to discontinue steroids prior to enrollment.
   2. Replacement doses, topical, ophthalmologic, and inhalational steroids are permitted.
5. History of CTCAE v5.0 Grade 4 immune-related AE due to adjuvant CTLA-4 or PD-1 blocking antibody.
6. Not fully recovered from adverse events (to Grade 1 or less [per CTCAE v5.0], with the exception of persistent alopecia, adrenal insufficiency, and hypothyroidism) due to prior treatment.
7. Active pneumonitis, history of pneumonitis that required steroids, or history of interstitial lung disease.
8. Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to poorly controlled hypertension, unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or greater), pericarditis within the previous 6 months, cerebrovascular accident, and implanted or continuous use of a pacemaker or defibrillator.
9. Known history of immunodeficiency.
10. Known additional malignancy that has progressed or required active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, curatively treated localized prostate cancer with prostate-specific antigen level below 4.0 ng/mL, in situ cervical cancer on biopsy or a squamous intraepithelial lesion on Papanicolaou smear, thyroid cancer (except anaplastic), and adjuvant hormonal therapy for breast cancer >3 years from curative-intent surgical resection.
11. Active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment.
12. Untreated, symptomatic, or enlarging central nervous system metastases or carcinomatous meningitis (including leptomeningeal metastases from solid tumors).
13. Prior allogenic tissue/solid organ transplant.
14. Known or suspected active infection with severe acute respiratory syndrome coronavirus 2 virus (SARS-CoV-2).
15. Active infection requiring systemic therapy.
16. Known or suspected infection with HIV, hepatitis B virus, or hepatitis C virus; testing is not required unless suspected.
17. Received a live/attenuated virus vaccination within 30 days prior to the first dose of study treatment on W1D1.
18. Received blood products (including platelets or red blood cells) or colony stimulating factors (including granulocyte colony stimulating factor, granulocyte/macrophage colony stimulating factor, or recombinant erythropoietin) within 30 days prior to the start of Screening.
19. History of allergy or hypersensitivity to nivolumab and/or any of its excipients.
20. Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the subject unable to cooperate or participate in the trial.
21. Participation in another clinical study of an investigational anticancer therapy or device within 30 days before the first dose of study treatment on W1D1.

    Note: Participation in the follow-up phase (receiving no study treatment) of a prior study is allowed.
22. Requires prohibited treatment (ie, non-protocol specified anticancer pharmacotherapy, surgery, or radiotherapy) for treatment of malignant tumor.
23. Has a life expectancy of less than 3 months and/or has rapidly progressing disease (eg, tumor bleeding, uncontrolled tumor pain) in the opinion of the treating Investigator.
24. Pregnant or breast-feeding or expecting to conceive or donate eggs within the projected duration of the study, from the time of consent until at least 150 days after the last dose of study treatment for women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (20):
- United States (20):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - California Cancer Associates for Research & Excellence, Inc., San Marcos, California
  - Hartford Healthcare, Hartford, Connecticut
  - Cleveland Clinic, Weston, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Louisville Health Care, Louisville, Kentucky
  - Atlantic Health, Morristown, New Jersey
  - Duke University Cancer Institute, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center / Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Texas Oncology, Sammons Cancer Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab Monotherapy: All participants received nivolumab monotherapy intravenously (IV) according to the treatment schedule.
- CMP-001 and Nivolumab: All participants received CMP-001 IT and nivolumab intravenously (IV) according to the treatment schedule.
Period: Overall Study
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Started (Received at least 1 dose of study treatment) | 11 | 9
Completed | 0 | 0
Not Completed | 11 | 9
Not completed — Sponsor Decision | 9 | 4
Not completed — Death | 2 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set (includes all participants who were randomized).
Groups:
- Nivolumab Monotherapy: All participants received nivolumab monotherapy IV according to the treatment schedule.
- CMP-001 and Nivolumab: All participants received CMP-001 IT and nivolumab IV according to the treatment schedule.
- Total: Total of all reporting groups
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (10.22) | 66.8 (7.14) | 69.3 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) by Blinded Independent Central Review (BICR)
Description: ORR, defined as the percentage of participants who have confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST vl.l) as assessed by Blinded Independent Central Review (BICR)
Time Frame: Up to approximately 39 months
Population: ITT Analysis Set (includes all participants who were randomized)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Percentage of participants | 73 [39.03 to 93.98] | 44 [13.70 to 78.80]

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Any Serious TEAE, and Any TEAE Leading to Discontinuation or Death
Description: Number of participants with any treatment-emergent adverse event (TEAE), any serious TEAE, and any TEAE leading to discontinuation or death reported.
Time Frame: Up to approximately 28 months (122 weeks)
Population: Safety Analysis Set (all participants who received at least 1 dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Participants
  Any TEAE | 11 | 9
  Any Serious TEAE | 5 | 2
  Any TEAE leading to death | 0 | 0

3. Secondary Outcome: Severity of TEAEs as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Description: Number of participants per NCI CTCAE version 5.0 Adverse Event Grade reported: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care activities of daily living; Grade 4 Life-threatening consequences: urgent intervention indicated; Grade 5 Death related to adverse event.
Time Frame: Up to approximately 28 months (122 weeks)
Population: Safety Analysis Set (all participants who received at least 1 dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Participants
  Grade 1 Mild | 2 | 0
  Grade 2 Moderate | 1 | 6
  Grade 3 Severe | 8 | 3
  Grade 4 Life-threatening | 0 | 0
  Grade 5 Death | 0 | 0

4. Secondary Outcome: Time to Response (TTR) by BICR
Description: TTR, defined as the time from the date of randomization to the first time when criteria are first met for complete response (CR) or partial response (PR), whichever occurred first, per RECIST vl.1 by BICR.
Time Frame: Up to approximately 39 months
Population: Number of participants analyzed for TTR included only participants in the ITT Analysis Set who had a confirmed best overall response (BOR) of CR or PR by BICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 8 | 4
Months | 2.14 [1.81 to 25.03] | 2.27 [2.07 to 4.70]

5. Secondary Outcome: Time to Response (TTR) by Investigator
Description: TTR, defined as the time from the date of randomization to the first time when criteria are first met for CR or PR, whichever occurred first, per RECIST vl.1 by Investigator.
Time Frame: Up to approximately 39 months
Population: Number of participants analyzed for TTR included only participants in the ITT Analysis Set who had a confirmed BOR of CR or PR by Investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 9 | 5
Months | 2.14 [1.81 to 3.48] | 3.45 [2.17 to 3.58]

6. Secondary Outcome: Duration of Response (DOR) by BICR
Description: DOR, defined as time from the date of first documented response (CR or PR) to the date of documented progressive disease (PD), based on RECIST vl.1 by BICR or death, whichever occurred first.
Time Frame: Up to approximately 39 months
Population: Number of participants analyzed for DOR included only participants in the ITT Analysis Set who had a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) by BICR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 8 | 4
Months | NA [NA to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated lower and upper confidence interval | NA [10.185 to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated upper confidence interval

7. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: DOR, defined as time from the date of first documented response (CR or PR) to the date of documented progressive disease (PD), based on RECIST vl.1 by Investigator or death, whichever occurred first.
Time Frame: Up to approximately 39 months
Population: Number of participants analyzed for DOR included only participants in the ITT Analysis Set who had a confirmed BOR of CR or PR by Investigator.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 9 | 5
Months | NA [4.172 to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated upper confidence interval | NA [6.702 to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated upper confidence interval

8. Secondary Outcome: Confirmed ORR in Non-injected Target Lesions by Investigator
Description: Confirmed ORR, defined as the percentage of participants in the analysis set who had confirmed BOR of CR or PR based on RECIST vl.1 as assessed by Investigator.
Time Frame: Up to approximately 39 months
Population: Number of participants analyzed included only participants in the ITT Analysis Set who had at least one non-injected target lesion, as assessed by Investigator, in the CMP-001 and Nivolumab reporting group, as prespecified by the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 and Nivolumab
Number analyzed (Participants) | 9
Percentage of participants | 56 [21.20 to 86.30]

9. Secondary Outcome: Progression-free Survival (PFS) by BICR
Description: PFS, defined as the time from the date of randomization to date of documented PD based on RECIST vl.1 by BICR or death, whichever occurred first.
Time Frame: Up to approximately 39 months
Population: ITT Analysis Set (includes all participants who were randomized)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Months | NA [2.070 to NA] — Median duration of PFS not reached; Insufficient number of participants with events for estimated upper confidence interval | 14.85 [1.971 to NA] — Insufficient number of participants with events for estimated upper confidence interval

10. Secondary Outcome: Progression-free Survival (PFS) by Investigator
Description: PFS, defined as the time from the date of randomization to date of documented PD based on RECIST vl.1 by Investigator or death, whichever occurred first.
Time Frame: Up to approximately 39 months
Population: ITT Analysis Set (includes all participants who were randomized)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Months | NA [2.103 to NA] — Median duration of PFS not reached; Insufficient number of participants with events for estimated upper confidence interval | 10.25 [1.971 to NA] — Insufficient number of participants with events for estimated upper confidence interval

11. Secondary Outcome: Overall Survival (OS) by Investigator
Description: OS, defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Up to approximately 40 months (174 weeks)
Population: ITT Analysis Set (includes all participants who were randomized)
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
Number analyzed (Participants) | 11 | 9
Months | NA [3.52 to 37.26] — Median duration of OS not reached | 20.04 [13.80 to 39.89]

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study up to approximately 40 months (174 weeks).
Arm/Group | Nivolumab Monotherapy | CMP-001 and Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/11 | 5/9
Serious Adverse Events (participants affected / at risk) | 5/11 | 2/9
Other Adverse Events (participants affected / at risk) | 11/11 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Monotherapy (N=11) | CMP-001 and Nivolumab (N=9)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Pseudomonal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Monotherapy (N=11) | CMP-001 and Nivolumab (N=9)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (13)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (8) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (6)
Chills (General disorders) | 1 (1) | 6 (47)
Fatigue (General disorders) | 5 (8) | 4 (9)
Pyrexia (General disorders) | 2 (2) | 3 (6)
Face oedema (General disorders) | 0 (0) | 1 (2)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site vesicles (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (6) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Achromotrichia acquired (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4)
Lipase increased (Investigations) | 2 (2) | 3 (6)
Weight decreased (Investigations) | 2 (3) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (2)
Activated partial thromboplastin time shortened (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (3)
Blood prolactin abnormal (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (11) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (6) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (5) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study stopped before reaching sample size as originally planned (n=140) for analysis per protocol. This was a business decision independent of safety/efficacy findings. Assessment of PK and immunotherapy was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04695977/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04695977/SAP_001.pdf